CLINICAL TRIAL: NCT01393327
Title: Feasibility and Influence of Respiratory and Exercise Therapy on Oxygen Uptake, Quality of Life and Right Heart Function in Chronic Thromboembolic Pulmonary Hypertension After Thromboendarterectomy
Brief Title: Feasibility and Influence of Exercise Therapy on Oxygen Uptake and Right Heart Function in CTEPH Patients After PEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S-488/2009
Record Dates: First submitted 2011-06-28; First posted 2011-07-13 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: CTEPH
Keywords: physical training; remaining post-operative pulmonary vascular changes; right ventricular pump function; PEA
MeSH Terms: interventions — Respiratory Rate; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory and exercise therapy (Experimental): Early after PEA postoperative three-week inpatient rehabilitation and subsequent continuing of the training at home for 12 weeks.
  Interventions: Behavioral: respiratory and exercise therapy

INTERVENTIONS:
Behavioral: respiratory and exercise therapy — Conventional therapy with diet, massage, relaxation baths, plus easy strolls specific respiratory and physical therapy plus mental walking training

SUMMARY:
Purpose of this study is to investigate whether and to what extent a cautious respiratory and movement therapy can complement medical treatment and the condition, oxygen uptake, quality of life, the pulmonary vascular pressures, the size of the right heart and the 6-minute walk distance in patients with pulmonary hypertension.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a complication of acute pulmonary embolism. According to current knowledge, it is caused by non-resolving fibrothrombotic obstructions of large pulmonary arteries. Some patients show an additional small vessel vasculopathy. Both kinds of obstruction lead to an increase in pulmonary vascular resistance (PVR), increase in mean pulmonary arterial pressure (mPAP), progressive right heart failure, and premature death if left untreated. Current guidelines recommend pulmonary endarterectomy (PEA) as the potentially curative treatment of first choice, which aims to remove fibrotic obstructions from the pulmonary vasculature. The survival of patients undergoing PEA surgery ranges between 76 and 91% after 3 years, which is superior to medical treatment in inoperable CTEPH patients. The majority of operated patients experience almost complete normalisation of haemodynamics and improvements in symptoms. However, 17-51% of operated patients will develop persistent or recurrent pulmonary hypertension (PH). Some patients remain limited in their exercise capacity and prognosis. As patients are monitored on an intensive care unit immediately after PEA, immobilisation after the operation may lead to further peripheral deconditioning. A recent study of 251 CTEPH patients with follow-up until 12 months after PEA showed a persistent exercise limitation in almost 40% of patients despite normalisation of PVR and haemodynamics. This limitation was characterised by a multifactorial aetiology also involving respiratory function abnormalities. Previous studies in patients with inoperable or persistent CTEPH have suggested beneficial effects of exercise training as an add-on to targeted medical therapy, increasing exercise capacity, and quality of life (QoL). However, it is not known, whether early rehabilitation with exercise treatment is safe, feasible, and may further improve exercise capacity after PEA. Prospective studies on exercise training for CTEPH patients shortly after PEA surgery are lacking. Furthermore, to the best of our knowledge, there have been no studies yet describing the early effect within the first weeks after PEA. The aim of this study was therefore to assess the feasibility of supervised exercise training in CTEPH patients shortly after PEA. Furthermore, changes of haemodynamic and clinical parameters including oxygen uptake, QoL, exercise capacity, and right heart function assessed by echocardiography and right heart catheterisation were obtained before and shortly after PEA.

ELIGIBILITY:
Inclusion Criteria:

* Consent form
* men and women> 18 years <80 years
* CTEPH after pulmonary endarterectomy

Exclusion Criteria:

* Patients with signs of right heart decompensation
* acute diseases, infections, fever
* Serious lung disease with FEV1 <50% or TLC <70% of target
* Other exclusion criteria are the following diseases: active myocarditis, unstable angina pectoris, exercise-induced ventricular arrhythmias, congestive heart failure, significant heart disease, pacemakers, and hypertrophic obstructive cardiomyopathy, or a highly reduced left ventricular function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Completion rate of exercise rehabilitation program training by CTEPH patients directly after PEA | up to 15 weeks after start of rehabilitation with exercise training
  Assessment of feasibility and tolerance of exercise rehabilitation directly after PEA assessed by the number of patients completing the exercise rehabilitation program
Change of peak O2 uptake (VO2peak) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Change of peak O2 uptake measured by cardiopulmonary exercise test (CPET)

SECONDARY OUTCOMES:
Change in right atrial pressure (RAP) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in right atrial pressure (RAP) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in right ventricular pressure (RVP) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in right ventricular pressure (RVP) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in systolic pulmonary arterial pressure (sPAP) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in systolic pulmonary arterial pressure (sPAP) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in diastolic pulmonary arterial pressure (dPAP) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in diastolic pulmonary arterial pressure (dPAP) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in mean pulmonary arterial pressure (mPAP) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in mean pulmonary arterial pressure (mPAP) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in pulmonary arterial wedge pressure (PAWP) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in pulmonary arterial wedge pressure (PAWP) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in cardiac output (CO) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in cardiac output (CO) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in pulmonary vascular resistance (PVR) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in pulmonary vascular resistance (PVR) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in venous oxygen saturation from pulmonary artery (SvO2) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in venous oxygen saturation from pulmonary artery (SvO2) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in cardiac index (CI) at rest | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics at rest
Change in cardiac index (CI) during exercise | up to 15 weeks after start of rehabilitation with exercise training
  Changes in hemodynamics during exercise
Change in exercise capacity assessed by six minute walking test | up to 15 weeks after start of rehabilitation with exercise training
  Six Minute Walking distance (6MWD) in meters
Change in exercise capacity - workload | up to 15 weeks after start of rehabilitation with exercise training
  recumbent bike (Workload in Watts) during cycle Ergometer test
Change in exercise capacity - respiratory economy | up to 15 weeks after start of rehabilitation with exercise training
  EqO2, EqCO2 assessed during cardiopulmonary exercise testing
Change of laboratory parameters of right heart function | up to 15 weeks after start of rehabilitation with exercise training
  Measurement of NT-proBNP
Change in right atrial area | up to 15 weeks after start of rehabilitation with exercise training
  Change of cm2 of right atrial area measured by 2D echocardiography
Change in right ventricular area | up to 15 weeks after start of rehabilitation with exercise training
  Change of cm2 of right ventricular area measured by 2D echocardiography
Change in visual right heart pump function | up to 15 weeks after start of rehabilitation with exercise training
  Change of category of right heart pump function (no impairment, slight impairment, moderate impairment, severe impairment) measured by 2D echocardiography
Safety of early rehabilitation directly after pulmonary endarterectomy: number of adverse events and serious adverse events | up to 15 weeks after start of rehabilitation with exercise training
  number of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, Professor, Study Director — Center for pulmonary hypertension, Thoraxclinic Heidelberg
Locations (1):
- Center for pulmonary Hypertension, Thoraxclinic Heidelberg, Heidelberg, Germany

REFERENCES:
- [Result] Delcroix M, Lang I, Pepke-Zaba J, Jansa P, D'Armini AM, Snijder R, Bresser P, Torbicki A, Mellemkjaer S, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Jais X, Ambroz D, Treacy C, Morsolini M, Jenkins D, Lindner J, Dartevelle P, Mayer E, Simonneau G. Long-Term Outcome of Patients With Chronic Thromboembolic Pulmonary Hypertension: Results From an International Prospective Registry. Circulation. 2016 Mar 1;133(9):859-71. doi: 10.1161/CIRCULATIONAHA.115.016522. Epub 2016 Jan 29. PMID 26826181
- [Result] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Result] Archibald CJ, Auger WR, Fedullo PF, Channick RN, Kerr KM, Jamieson SW, Kapelanski DP, Watt CN, Moser KM. Long-term outcome after pulmonary thromboendarterectomy. Am J Respir Crit Care Med. 1999 Aug;160(2):523-8. doi: 10.1164/ajrccm.160.2.9808109. PMID 10430723
- [Result] Condliffe R, Kiely DG, Gibbs JS, Corris PA, Peacock AJ, Jenkins DP, Hodgkins D, Goldsmith K, Hughes RJ, Sheares K, Tsui SS, Armstrong IJ, Torpy C, Crackett R, Carlin CM, Das C, Coghlan JG, Pepke-Zaba J. Improved outcomes in medically and surgically treated chronic thromboembolic pulmonary hypertension. Am J Respir Crit Care Med. 2008 May 15;177(10):1122-7. doi: 10.1164/rccm.200712-1841OC. Epub 2008 Feb 21. PMID 18292468
- [Result] Skoro-Sajer N, Marta G, Gerges C, Hlavin G, Nierlich P, Taghavi S, Sadushi-Kolici R, Klepetko W, Lang IM. Surgical specimens, haemodynamics and long-term outcomes after pulmonary endarterectomy. Thorax. 2014 Feb;69(2):116-22. doi: 10.1136/thoraxjnl-2013-203746. Epub 2013 Sep 19. PMID 24052543
- [Result] Matsuda H, Ogino H, Minatoya K, Sasaki H, Nakanishi N, Kyotani S, Kobayashi J, Yagihara T, Kitamura S. Long-term recovery of exercise ability after pulmonary endarterectomy for chronic thromboembolic pulmonary hypertension. Ann Thorac Surg. 2006 Oct;82(4):1338-43; discussion 1343. doi: 10.1016/j.athoracsur.2006.03.105. PMID 16996930
- [Result] Wieteska M, Biederman A, Kurzyna M, Dyk W, Burakowski J, Wawrzynska L, Szturmowicz M, Fijalkowska A, Szatkowski P, Torbicki A. Outcome of Medically Versus Surgically Treated Patients With Chronic Thromboembolic Pulmonary Hypertension. Clin Appl Thromb Hemost. 2016 Jan;22(1):92-9. doi: 10.1177/1076029614536604. Epub 2014 May 28. PMID 24875780
- [Result] Simonneau G, D'Armini AM, Ghofrani HA, Grimminger F, Hoeper MM, Jansa P, Kim NH, Wang C, Wilkins MR, Fritsch A, Davie N, Colorado P, Mayer E. Riociguat for the treatment of chronic thromboembolic pulmonary hypertension: a long-term extension study (CHEST-2). Eur Respir J. 2015 May;45(5):1293-302. doi: 10.1183/09031936.00087114. Epub 2014 Nov 13. PMID 25395036
- [Result] Fukui S, Ogo T, Goto Y, Ueda J, Tsuji A, Sanda Y, Kumasaka R, Arakawa T, Nakanishi M, Fukuda T, Takaki H, Yasuda S, Ogawa H, Nakanishi N. Exercise intolerance and ventilatory inefficiency improve early after balloon pulmonary angioplasty in patients with inoperable chronic thromboembolic pulmonary hypertension. Int J Cardiol. 2015 Feb 1;180:66-8. doi: 10.1016/j.ijcard.2014.11.187. Epub 2014 Nov 26. No abstract available. PMID 25438215
- [Result] Corsico AG, D'Armini AM, Conio V, Sciortino A, Pin M, Grazioli V, Di Vincenzo G, Di Domenica R, Celentano A, Vanini B, Grosso A, Gini E, Albicini F, Merli VN, Ronzoni V, Ghio S, Klersy C, Cerveri I. Persistent exercise limitation after successful pulmonary endoarterectomy: frequency and determinants. Respir Res. 2019 Feb 14;20(1):34. doi: 10.1186/s12931-019-1002-5. PMID 30764853
- [Result] Ehlken N, Lichtblau M, Klose H, Weidenhammer J, Fischer C, Nechwatal R, Uiker S, Halank M, Olsson K, Seeger W, Gall H, Rosenkranz S, Wilkens H, Mertens D, Seyfarth HJ, Opitz C, Ulrich S, Egenlauf B, Grunig E. Exercise training improves peak oxygen consumption and haemodynamics in patients with severe pulmonary arterial hypertension and inoperable chronic thrombo-embolic pulmonary hypertension: a prospective, randomized, controlled trial. Eur Heart J. 2016 Jan 1;37(1):35-44. doi: 10.1093/eurheartj/ehv337. Epub 2015 Jul 31. PMID 26231884
- [Result] Grunig E, Lichtblau M, Ehlken N, Ghofrani HA, Reichenberger F, Staehler G, Halank M, Fischer C, Seyfarth HJ, Klose H, Meyer A, Sorichter S, Wilkens H, Rosenkranz S, Opitz C, Leuchte H, Karger G, Speich R, Nagel C. Safety and efficacy of exercise training in various forms of pulmonary hypertension. Eur Respir J. 2012 Jul;40(1):84-92. doi: 10.1183/09031936.00123711. Epub 2012 Feb 9. PMID 22323570
- [Result] Lankeit M, Krieg V, Hobohm L, Kolmel S, Liebetrau C, Konstantinides S, Hamm CW, Mayer E, Wiedenroth CB, Guth S. Pulmonary endarterectomy in chronic thromboembolic pulmonary hypertension. J Heart Lung Transplant. 2017 Jul 1:S1053-2498(17)31877-6. doi: 10.1016/j.healun.2017.06.011. Online ahead of print. PMID 28750932
- [Result] Kovacs G, Avian A, Pienn M, Naeije R, Olschewski H. Reading pulmonary vascular pressure tracings. How to handle the problems of zero leveling and respiratory swings. Am J Respir Crit Care Med. 2014 Aug 1;190(3):252-7. doi: 10.1164/rccm.201402-0269PP. PMID 24869464
- [Result] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Result] Grunig E, Biskupek J, D'Andrea A, Ehlken N, Egenlauf B, Weidenhammer J, Marra AM, Cittadini A, Fischer C, Bossone E. Reference ranges for and determinants of right ventricular area in healthy adults by two-dimensional echocardiography. Respiration. 2015;89(4):284-93. doi: 10.1159/000371472. Epub 2015 Mar 7. PMID 25765954
- [Result] Grunig E, Henn P, D'Andrea A, Claussen M, Ehlken N, Maier F, Naeije R, Nagel C, Prange F, Weidenhammer J, Fischer C, Bossone E. Reference values for and determinants of right atrial area in healthy adults by 2-dimensional echocardiography. Circ Cardiovasc Imaging. 2013 Jan 1;6(1):117-24. doi: 10.1161/CIRCIMAGING.112.978031. Epub 2012 Nov 29. PMID 23197080
- [Result] Leung Wai Sang S, Morin JF, Hirsch A. Operative and Functional Outcome After Pulmonary Endarterectomy for Advanced Thromboembolic Pulmonary Hypertension. J Card Surg. 2016 Jan;31(1):3-8. doi: 10.1111/jocs.12646. Epub 2015 Nov 4. PMID 26537658
- [Result] Li YD, Zhai ZG, Wu YF, Yang YH, Gu S, Liu Y, Su PX, Wang C. Improvement of right ventricular dysfunction after pulmonary endarterectomy in patients with chronic thromboembolic pulmonary hypertension: utility of echocardiography to demonstrate restoration of the right ventricle during 2-year follow-up. Thromb Res. 2013 May;131(5):e196-201. doi: 10.1016/j.thromres.2013.02.001. Epub 2013 Feb 27. PMID 23453712
- [Result] Raza F, Vaidya A, Lacharite-Roberge AS, Lakhter V, Al-Maluli H, Ahsan I, Boodram P, Dass C, Rogers F, Keane MG, Weaver S, Bashir R, Toyoda Y, Forfia P. Initial clinical and hemodynamic results of a regional pulmonary thromboendarterectomy program. J Cardiovasc Surg (Torino). 2018 Jun;59(3):428-437. doi: 10.23736/S0021-9509.17.10188-6. Epub 2017 Sep 4. PMID 28870062
- [Result] Kepez A, Sunbul M, Kivrak T, Eroglu E, Ozben B, Yildizeli B, Mutlu B. Evaluation of improvement in exercise capacity after pulmonary endarterectomy in patients with chronic thromboembolic pulmonary hypertension: correlation with echocardiographic parameters. Thorac Cardiovasc Surg. 2014 Feb;62(1):60-5. doi: 10.1055/s-0033-1336012. Epub 2013 Apr 5. PMID 23564536
- [Result] La Rovere MT, Pinna GD, Pin M, Bruschi C, Callegari G, Zanotti E, D'Armini A, Ambrosino N. Exercise Training After Pulmonary Endarterectomy for Patients with Chronic Thromboembolic Pulmonary Hypertension. Respiration. 2019;97(3):234-241. doi: 10.1159/000492754. Epub 2018 Oct 5. PMID 30293071
- [Result] Guth S, Wiedenroth CB, Rieth A, Richter MJ, Gruenig E, Ghofrani HA, Arlt M, Liebetrau C, Prufer D, Rolf A, Hamm CW, Mayer E. Exercise right heart catheterisation before and after pulmonary endarterectomy in patients with chronic thromboembolic disease. Eur Respir J. 2018 Sep 17;52(3):1800458. doi: 10.1183/13993003.00458-2018. Print 2018 Sep. PMID 30139773
- [Result] Adams V, Reich B, Uhlemann M, Niebauer J. Molecular effects of exercise training in patients with cardiovascular disease: focus on skeletal muscle, endothelium, and myocardium. Am J Physiol Heart Circ Physiol. 2017 Jul 1;313(1):H72-H88. doi: 10.1152/ajpheart.00470.2016. Epub 2017 May 5. PMID 28476924
- [Result] Pearson MJ, Smart NA. Exercise therapy and autonomic function in heart failure patients: a systematic review and meta-analysis. Heart Fail Rev. 2018 Jan;23(1):91-108. doi: 10.1007/s10741-017-9662-z. PMID 29185161
- [Result] Paneroni M, Simonelli C, Vitacca M, Ambrosino N. Aerobic Exercise Training in Very Severe Chronic Obstructive Pulmonary Disease: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2017 Aug;96(8):541-548. doi: 10.1097/PHM.0000000000000667. PMID 28099192
- [Result] Piepoli MF. Exercise training in chronic heart failure: mechanisms and therapies. Neth Heart J. 2013 Feb;21(2):85-90. doi: 10.1007/s12471-012-0367-6. PMID 23239451
- [Result] Anderson L, Nguyen TT, Dall CH, Burgess L, Bridges C, Taylor RS. Exercise-based cardiac rehabilitation in heart transplant recipients. Cochrane Database Syst Rev. 2017 Apr 4;4(4):CD012264. doi: 10.1002/14651858.CD012264.pub2. PMID 28375548
- [Derived] Nagel C, Nasereddin M, Benjamin N, Egenlauf B, Harutyunova S, Eichstaedt CA, Xanthouli P, Mayer E, Grunig E, Guth S. Supervised Exercise Training in Patients with Chronic Thromboembolic Pulmonary Hypertension as Early Follow-Up Treatment after Pulmonary Endarterectomy: A Prospective Cohort Study. Respiration. 2020;99(7):577-588. doi: 10.1159/000508754. Epub 2020 Jul 29. PMID 32726793